CLINICAL TRIAL: NCT04552158
Title: Nutritional Assessment and Impact of the Mediterranean Diet on Patients With Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yasmin Ashraf Mahmoud Osman (Other)
Responsible Party: Sponsor-Investigator, Yasmin Ashraf Mahmoud Osman, assistant lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: nutrition and IBD
Record Dates: First submitted 2020-09-06; First posted 2020-09-17 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2020-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: All Patients will be subjected to assessment of their nutritional status at day 0 and after 3 months of only medical management for the control group and of combined medical and nutritional management using Mediterranean dietary pattern for the experimental group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controlled group (No Intervention): patients with IBD who will be assessed for their nutritional status at day 0 and after 3 months of medical management only
- experimental group (Experimental): patients with IBD who will be assessed for their nutritional status at day 0 and after 3 months of medical management and nutritional management in the form of the Mediterranean diet
  Interventions: Dietary Supplement: Mediterranean diet

INTERVENTIONS:
Dietary Supplement: Mediterranean diet — The Mediterranean diet (MedDiet) is a nutritional model inspired by the traditional dietary pattern of some of the countries of the Mediterranean basin. Mediterranean dietary pattern (MDP) gather the following characteristics: abundant consumption of olive oil and high consumption of fruits, vegetables, cereals (preferably as whole grain), legumes, nuts and seeds. The MDP also includes moderate consumption of fish and shellfish, white meat, eggs, and fermented dairy products (cheese and yogurt), as well as relatively small amounts of red meat, processed meats, and foods rich in sugars. Frequent but moderate intake of wine, especially red wine with meals is also recommended
  Arms: experimental group

SUMMARY:
1. Assessment of nutritional status among patients with inflammatory bowel disease using different nutritional assessment tools.
2. Assessment of correlation between nutritional status and disease severity.
3. Assessment of the impact of the Mediterranean diet on the nutritional status of the patients after 3 months.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) comprise a variety of disorders that result from the continuous activation of the immunoinflammatory cascade, whose etiology has not been defined in some cases. Classical IBD include Crohn's disease (CD), ulcerative colitis (UC), and indeterminate colitis. These diseases are chronic and are characterized by alternating periods of recurrence and remission.

The European Society of Clinical Nutrition and Metabolism (ESPEN) defined malnutrition as a state resulting from lack of uptake or intake of nutrition leading to altered body composition (decreased fat-free mass and body cell mass), resulting in diminished physical and mental function and impaired clinical outcome from disease.

The prevalence of Malnutrition in patients with inflammatory bowel disease (IBD) is very high. it presents in up to 70% of patients with active disease and up to 38% in patients with remission.

Several factors contribute to the malnutrition in IBD including insufficient nutrient intake as a consequence of impaired appetite (anorexia, stomachache), short bowel syndrome, impaired nutrient absorption (diarrhea, villus atrophy, bowel resection, intestinal flora overgrowth), increased nutrient losses (bleeding, fistulae), and food-drug interaction.

Malnutrition in IBD has been associated with several adverse clinical outcomes. IBD patients with nutritional deficiencies may present with higher mortality rate, length of stay in the hospital, infectious rate, and even thromboembolic events than those without nutritional deficiencies. Furthermore, undernutrition in patients with postoperative conditions has been associated with increased complications such as anastomotic leakage and breakdown, infection including sepsis and pneumonia, prolonged hospitalization, and increased mortality.

IBD is clearly associated with intestinal dysbiosis. Changes in the microbiome have a pivotal role in determining the onset of the pathology, when the genetic background of the individual makes him/her predisposed and other concomitant environmental factors intervene. Results of studies aimed at characterizing the microbiota of patients suffering from IBD, even sometimes with checkered results, indicate a generalized decrease in biodiversity, measured by an appropriate parameter-alpha-as well as a reduction in specific taxa including Firmicutes and Bacteroidetes, Lactobacillus and Eubacterium. IBD patients also present a reduction in species producing butyrate, a short chain fatty acid positively modulating intestinal homeostasis and reducing inflammation.

Regarding environmental factors, accumulating data have proven that various nutritional components in diet can play a significant role in the development and clinical course of IBD. Dietary nutrients alter the composition of the gut microbiota and intestinal permeability, influencing the interaction between the host and gut microbiota.

The Mediterranean diet (MedDiet) is a nutritional model inspired by the traditional dietary pattern of some of the countries of the Mediterranean basin. Mediterranean dietary pattern (MDP) gather the following characteristics: abundant consumption of olive oil and high consumption of fruits, vegetables, cereals (preferably as whole grain), legumes, nuts and seeds. The MDP also includes moderate consumption of fish and shellfish, white meat, eggs, and fermented dairy products (cheese and yogurt), as well as relatively small amounts of red meat, processed meats, and foods rich in sugars. Frequent but moderate intake of wine, especially red wine with meals is also recommended.

Results from clinical and translational research on the Mediterranean diet point to its possible meaningful use in managing IBD, and thus additional studies could have the potential to add further insights to the field. Concerning published data, it was observed that 153 Italian healthy subjects were investigated for their dietary habits and their gut microbiota was assessed, and high-level adherence to a Mediterranean diet was found to beneficially impact the gut microbiota and associated metabolome. These studies provided the first concrete evidence for the interconnection between Mediterranean dietary patterns, gut microbiota and microbial metabolites as they observed that the consumption of fruit, vegetables and legumes by subjects with satisfactory adherence to the Mediterranean diet was associated with an increase in fecal SCFA levels, an effect that was likely boosted by bacteria belonging to both the Firmicutes and Bacteroidetes capable of degrading carbohydrates not digestible by the host. When eight adult patients suffering from CD followed the Mediterranean diet for 6 weeks, their transcriptome analysis showed a change in expression of more than 3000 genes; changes in the intestinal microbiota, although not significant, showed a trend towards normalization with an increase in the expression of Bacteroidetes (17.89% to 18.74%), Clostridium cluster IV (19.2% to 21.86%) and Clostridium cluster XIVa (26.78% to 28.79%) and a decrease in the abundance of Proteobacteria (5.93% to 5.48%) and Bacillaceae (4.65% to 4.21%).

ELIGIBILITY:
Inclusion Criteria:

* patients with inflammatory bowel disease between 18 to 55 years

Exclusion Criteria:

* presence of other diseases that affect the nutritional status of the patients like diabetes mellitus, liver cirrhosis, chronic kidney disease, and malignancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of nutritional status among patients with inflammatory bowel disease using body weight | Two time points: Change in body weight at patient presentation and after 3 months of medical management only
  current body weight in kilograms will be measured
Assessment of nutritional status among patients with inflammatory bowel disease using body mass index (BMI) | Two time points: Change in BMI at patient presentation and after 3 months of medical management only
  current body weight in kilograms and height in meters will be measured BMI is calculated in kg/m2
Assessment of nutritional status among patients with inflammatory bowel disease using the anthropometric measures | Two time points: Change in the anthropometric parameters at patient presentation and after 3 months of medical management only
  triceps skin fold thickness (TST) in mm, mid arm circumference(MAC) in cm and mid arm muscle circumference in cm (MAMC) MAMC (cm) = MAC(cm) - { 0.314 X TST(mm) }.
Assessment of nutritional status among patients with inflammatory bowel disease using prognostic nutritional index (PNI) | Two time points: Change in PNI score at patient presentation and after 3 months of medical management only
  prognostic nutritional index (PNI) which is score derived from total lymphocytic count (TLC)and serum albumin (PNI = albumin g/dl x 10 + TLC/µL x 0.005)
Assessment of nutritional status among patients with inflammatory bowel disease using controlling nutritional status(CONUT) | Two time points: Change in CONUT score at patient presentation and after 3 months of medical management only
  controlling nutritional status (CONUT) is also a score derived from total lymphocytic count, serum albumin and blood cholesterol level

SECONDARY OUTCOMES:
Assessment of the impact of Mediterranean diet on the nutritional status for patients who received the Mediterranean diet after 3 months | after 3 months of medical and Mediterranean diet management
  This assessment is based on an individualised scoring system of 7 points for the measured nutritional parameters, in which patients who have > 3 points are considered to have a better outcome.

REFERENCES:
- [Background] Lee D, Albenberg L, Compher C, Baldassano R, Piccoli D, Lewis JD, Wu GD. Diet in the pathogenesis and treatment of inflammatory bowel diseases. Gastroenterology. 2015 May;148(6):1087-106. doi: 10.1053/j.gastro.2015.01.007. Epub 2015 Jan 15. PMID 25597840
- [Background] Lane ER, Zisman TL, Suskind DL. The microbiota in inflammatory bowel disease: current and therapeutic insights. J Inflamm Res. 2017 Jun 10;10:63-73. doi: 10.2147/JIR.S116088. eCollection 2017. PMID 28652796
- [Background] Weber AT, Shah ND, Sauk J, Limketkai BN. Popular Diet Trends for Inflammatory Bowel Diseases: Claims and Evidence. Curr Treat Options Gastroenterol. 2019 Dec;17(4):564-576. doi: 10.1007/s11938-019-00248-z. PMID 31705371